CLINICAL TRIAL: NCT00712686
Title: A Multicenter, Double-Blind, Randomized, Comparative Study of Aripiprazole and Olanzapine in the Treatment of Patients With Acute Schizophrenia
Brief Title: Comparative Study of Aripiprazole and Olanzapine in the Treatment of Patients With Acute Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-003
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2010-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- B1 (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 15-30 mg, once daily, 140 weeks
  Other Names: Abilify
  Arms: A1
Drug: Olanzapine — Capsule, Oral, 10-20 mg, once daily, 140 weeks
  Arms: B1

SUMMARY:
The purpose of this study is to compare the efficacy and tolerability of aripiprazole to olanzapine over 26 weeks for the treatment of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Patients with DSM-IV diagnosis of schizophrenia patients in acute relapse
* Treated as outpatients for at least one continuous 3-month period during the past 12 months
* PANSS total score ≥60
* Previously responsive to neuroleptics (other than clozapine)
* Able to give informed consent and comprehend and satisfactorily comply with the protocol requirements

Exclusion Criteria:

* An Axis I (DSM-IV) diagnosis of schizoaffective disorder
* A clinical picture and/or history that was consistent with: (a) Delirium, dementia, amnestic or other cognitive disorders; (b) Bipolar disorder; (c)personality disorder
* Nonresponsive to prior olanzapine therapy
* Likely to require prohibited concomitant therapy
* DSM-IV criteria for any significant substance abuse within the past three months, including addiction to cocaine or alcohol
* Known to be allergic or hypersensitive to study drugs
* Represented a significant risk of committing suicide based on history or mental status exam
* Unstable thyroid pathology and treatment within the past six months
* A history or evidence of a medical condition that would expose the patient to an undue risk
* Clinically significant abnormal laboratory test results (including urine drug screen), vital sign, or ECG findings

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2000-06; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
The mean change in the PANSS Total Score | from baseline to Week 6
The percentage of patients showing significant weight gain (a≥ 7% increase) | from baseline to Week 26

SECONDARY OUTCOMES:
Change from baseline on the CGI-S Score | at the end of study
Change from baseline on PANSS Total Score | at the end of study
Change from baseline on PANSS-Positive Scale Total Score | at the end of study
Change from baseline on PANSS-Negative Scale Total Score | at the end of study
Mean change from baseline in PANSS-derived Brief Psychiatric Rating Scale (BPRS) Core Score | at the end of study
Mean CGI-I Score | at the end of study
Percentage of responders (≥ 30% decrease in PANSS Total Score, or score of 1 or 2 on CGI-I) | at the end of study
Change from baseline on the MADRS | at the end of study
Safety and tolerability | at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Background] Fleischhacker WW, McQuade RD, Marcus RN, Archibald D, Swanink R, Carson WH. A double-blind, randomized comparative study of aripiprazole and olanzapine in patients with schizophrenia. Biol Psychiatry. 2009 Mar 15;65(6):510-7. doi: 10.1016/j.biopsych.2008.07.033. Epub 2008 Nov 4. PMID 18986646